CLINICAL TRIAL: NCT03140748
Title: Kinetics of Serum β-D-glucan During Peritonitis With Candida in Resuscitation
Acronym: PERIGLUC1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PI2016_843_0036
Record Dates: First submitted 2017-04-14; First posted 2017-05-04 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Peritonitis Infectious; Candida Infection
MeSH Terms: conditions — Candidiasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with fungal peritonitis (Other)
  Interventions: Other: To evaluate the initial levels and kinetics of serum β-D-glucan
- Patients with peritonitis without yeast (Other)
  Interventions: Other: To evaluate the initial levels and kinetics of serum β-D-glucan

INTERVENTIONS:
Other: To evaluate the initial levels and kinetics of serum β-D-glucan — To evaluate the initial levels and kinetics of serum β-D-glucan during fungal peritonitis compared to a control group of yeast-free peritonitis

SUMMARY:
Intraabdominal fungal infections with Candida are constantly increasing. Their diagnosis and treatment is difficult. Morbidity and mortality are high. Β-D-Glucan has been proposed as a marker of systemic fungal infection in candidemia. Moreover, its kinetics is associated with therapeutic success. On the other hand, there are no data on intraabdominal infections that are much more frequent. The objective of the study is to evaluate the initial levels of β-D-glucan and its daily kinetics during the treatment of fungal peritonitis in resuscitation compared to a control group with a yeast-free peritonitis.

ELIGIBILITY:
Inclusion Criteria:

* Major Patient (age ≥ 18 years)
* Community or associated peritonitis, operated and hospitalized in resuscitation
* Affiliation to a social security scheme

Exclusion Criteria:

* Allergy known to echinocandins
* Dying Patient
* Limitation of care
* Predictable duration of follow-up ≤ 10 days
* Transfusion within 3 months
* Patient minor, patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-08-22 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Blood determination of serum β-D-glucan kinetics in patients with peritonitis | 28 days
  Blood determination of serum β-D-glucan kinetics in patients with peritonitis

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

REFERENCES:
- [Result] Dupont H, Malaquin S, Villeret L, Macq PY, Ammenouche N, Tinturier F, Diouf M, Rumbach M, Chouaki T. Is ss-d-glucan Relevant for the Diagnosis and Follow-Up of Intensive Care Patients with Yeast-Complicated Intra-Abdominal Infection? J Fungi (Basel). 2022 May 6;8(5):487. doi: 10.3390/jof8050487. PMID 35628743